CLINICAL TRIAL: NCT07192588
Title: A Randomised, Double-Blind, Vehicle-Controlled, Multi-Centre, Parallel-Group Study to Investigate the Safety, Tolerability, and Efficacy of GR1014 Cutaneous Gel as a Topical Radioprotector in the Prevention of the Radiodermatitis Occurring With Adjuvant Radiotherapy for Localised Breast Cancer After Lumpectomy
Brief Title: A Study of GR1014 Cutaneous Gel for the Prevention of Skin Reactions Caused by Radiation Therapy for Breast Cancer
Acronym: GuARD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Graegis Pharmaceuticals Ltd (Industry)
Collaborators: Excelya (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GRA.05.SPR.0001; 2023-508728-36-00 (EU CTIS Number); 1009515 (Other: MHRA (IRAS number))
Record Dates: First submitted 2025-09-11; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Radiodermatitis; Acute
Keywords: Radiotherapy; Amifostine thiol; Radiodermatitis; Prevention; Cutaneous; Breast Cancer; Topical
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GR1014-CG 4.7% (Experimental): GR1014-CG 4.7% will be applied topically on the breast skin surface to be irradiated 15-30 min each day of the radiotherapy, 15-30 min before irradiation
  Interventions: Radiation: Radiation Therapy; Drug: GR1014-CG 4.7%
- GR1014-CG 2.4% (Experimental): GR1014-CG 2.4% will be applied topically on the breast skin surface to be irradiated 15-30 min each day of the radiotherapy, 15-30 min before irradiation
  Interventions: Drug: GR1014-CG 2.4%; Radiation: Radiation Therapy
- Vehicle Gel (Placebo Comparator): Vehicle Gel will be applied topically on the breast skin surface to be irradiated 15-30 min each day of the radiotherapy, 15-30 min before irradiation
  Interventions: Drug: Vehicle Gel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: GR1014-CG 2.4% — Topical gel formulation of amifostine thiol (GR1014) at 25 mg/mL
  Arms: GR1014-CG 2.4%
Drug: Vehicle Gel — The same topical formulation as GR1014-CG without the active ingredient amifostine thiol
  Arms: Vehicle Gel
Radiation: Radiation Therapy — Ultra hypofractionated RT, 26 Gy in 5 daily fractions (5.2 Gy) given over 1 week on the whole breast
Drug: GR1014-CG 4.7% — Topical gel formulation of amifostine thiol (GR1014) at 50 mg/mL
  Arms: GR1014-CG 4.7%

SUMMARY:
This clinical trial is testing a new skin gel called GR1014-CG to evaluate its safety and see if it can help prevent or reduce skin irritation (such as redness, soreness, etc.) caused by radiation therapy (RT) after breast-conserving surgery for early-stage breast cancer. The study is for women aged 18 and older who have had surgery to remove a breast tumor and need radiation therapy.

The main goals of the study are to find out:

* If GR1014-CG is safe to use
* If the gel can prevent or lower the severity of skin irritation caused by RT.

During the study participants will,

* Be randomly assigned to use one of two strengths of GR1014-CG (4.7% or 2.4%) or a placebo gel (a gel with no active drug).
* Apply the gel to the breast before each radiation session for 5 days.
* Visit the clinic once a week for 4 weeks to check their skin and overall health. At the end of the 4th week, if there are still signs of irritation participants will come to the clinic for a checkup 2 weeks after, and then again 2 weeks after if the irritation is still observed.
* Keep a diary to record any pain or itching they may feel.

DETAILED DESCRIPTION:
Adjuvant radiation therapy (RT) decreases the chances of local cancer reappearance and improves survival rates. However, radiotherapy is often associated with side effects, including radiation-induced dermatitis (radiodermatitis). Symptoms of radiation-induced dermatitis include skin redness (erythema), swelling (oedema), dry or moist peeling of the skin (desquamation), and varying degrees of pain. GR1014 cutaneous gel (GR1014-CG) contains amifostine thiol (GR1014), an active substance with well-established radioprotective effects. The protective properties of GR1014-CG are potentially beneficial in preventing radiodermatitis, particularly in patients with breast cancer treated with adjuvant RT. GR1014 CG is designed to be topically applied to the skin before each RT session without any modifications to the planned course of RT.

This is a dose-finding, phase-2 trial to investigate the safety, tolerability, and efficacy of GR1014-CG as a topical radioprotector in the reduction of radiodermatitis occurring in patients treated with adjuvant ultra-hypofractionated RT (26 Gy in 5 fractions over 1 week) for localized, non-metastatic breast cancer after tumor removal (lumpectomy) versus vehicle gel.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age ≥18 years. Those of childbearing potential must be using highly effective contraception methods during the study and for 30 days after the last administration of the study treatment and have a negative pregnancy test at screening and no more than 10 days prior to the administration of the first dose of study treatment
* Patients with primary, localized breast cancer without metastases pTis, T1-3, pN0-N1mi, M0, who have undergone breast-conserving surgical excision and require adjuvant RT. The patients should be randomized after having recovered from the last surgery and, if delivered, the adjuvant chemotherapy. The patients can be included no matter the status of estrogen and progesterone receptors, malignancy grade, or HER2 status.
* ECOG performance status 0-2
* Patients to be treated with ultra hypofractionated RT, 26 Gy in 5 fractions (5.2 Gy) on whole breast (EQD2 > 42.6 Gy for α/β of 3)
* Patients with no signs of dermatitis in the breast area to be irradiated, i.e., assessed Grade 0 as per CTCAE radiation dermatitis grading
* Patients whom the investigator has deemed able to comply with the RT and investigational treatment done under the supervision of the medical personnel throughout the study period
* Patients who have completed the appropriate washout period for any prior interventions or treatments

Exclusion Criteria:

* Pregnant and breastfeeding women
* Patients under any treatment concomitant to radiotherapy tested in another clinical study
* Allergies to any of the ingredients in GR1014-CG
* Patients protected by law (legal guardianship or protection)
* Patients unable to adhere to the requirements of the study
* History of thoracic RT
* Participants with the presence of skin rash, ulceration, unhealed surgical wounds, biopsy sites, or open wound in the breast or chest area at visit 2
* Patients suffering from scleroderma, auto-immune disease, micro-vascular diseases, collagen tissue diseases, lupus, pre-existing loss of skin integrity, active eczema in the region to be treated or with a history of any of the following: drug-induced severe cutaneous adverse reaction (SCAR; including, but not limited to Stevens-Johnson syndrome/toxic epidermal necrolysis [SJS/TEN], or drug reaction with eosinophilia and systemic symptoms)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with No Radiation Dermatitis as Assessed by CTCAE Latest Version (LV) (Grade of 0) | At any time between the first radiotherapy session and 4 weeks after the last one
  As per CTCAE - Radiation Dermatitis: A finding of cutaneous inflammatory reaction occurring as a result of exposure to biologically effective levels of ionizing radiation.
  Grade 1: Faint erythema or dry desquamation; Grade 2: Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin folds and creases; moderate edema; Grade 3: Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion; Grade 4: Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated; Grade 5: Death

SECONDARY OUTCOMES:
Percentage of Participants with a Radiodermatitis grade ≥2 (CTCAE LV) | At any time between the first radiotherapy session and 4 weeks after the last one
Percentage of Participants with No Radiation Dermatitis (CTCAE LV) | 4 weeks after the last radiotherapy session (at Visit 10)
Maximum Grade of Radiodermatitis (CTCAE LV) Reached in each Participant | Between the first radiotherapy session and 4 weeks after the last one
Assessments of Radiodermatitis Grade (CTCAE LV) | Between the first radiotherapy session and up to 8 weeks after the last one
Time to Onset of Radiodermatitis Grade ≥2 (CTCAE LV). | From the first radiotherapy session and up to 8 weeks after the last one
Duration of Radiodermatitis Grade ≥2 (CTCAE LV) | From the first session of radiotherapy and up to 8 weeks after the last one
Percentage of participants with severe radiodermatitis (grade ≥3; CTCAE LV) | At any time between the first radiotherapy session and 4 weeks after the last one
Number of cases of side effects of radiotherapy other than radiodermatitis | At any time between the first radiotherapy session and up to 8 weeks after the last one
  Oedema; hyperpigmentation; skin infection; need for topical and systemic antibiotics; need for topical steroids; need for analgesics; need for silicone-based dressings
Absolute change from baseline in weekly averaged worst skin pain score in the irradiated area | From date of screening visit and up to 8 weeks after the last radiotherapy session
  Worst pain intensity (during the last 24 hours) will be scored daily on a 0-10 Numeric Rating Scale. Zero is equivalent to no pain and 10 indicates the worst possible pain
Absolute change from baseline in weekly averaged peak pruritus score in the irradiated area. | From date of screening visit and up to 8 weeks after the last radiotherapy session
  Peak pruritus intensity (during the last 24 hours) scored daily on a 0-10 NRS. Zero is equivalent to no pruritus (itching) and 10 indicates the worst possible pruritus.
Total score and sub-scores of Dermatology Life Quality Index (DLQI) | From the first radiotherapy session and up to 8 weeks after the last one
  DLQI is a ten-item questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. There are 10 questions covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- The Royal Marsden NHS Foundation Trust and The Institute of Cancer Research, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No